CLINICAL TRIAL: NCT06451874
Title: Motoric Cognitive Risk Syndrome: Refining Treatment Strategies and Testing Feasibility to Personalize Treatment for Older Veterans
Brief Title: Personalized Exercise Treatments for Older Veterans With Motoric Cognitive Risk Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: E5294-W
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Motoric Cognitive Risk Syndrome
Keywords: Veterans; Mobility; Cognition; Sequential Multiple Assignment Randomized Trial

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial (SMART)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage 1 Exercise Treatment (Experimental): Participants will first be randomized to 6-week exercise treatment (FPT or MBDT)
  Interventions: Behavioral: Functional Power Training (FPT); Behavioral: Music-Based Digital Therapy (MBDT)
- Stage 2: Exercise Treatment (Experimental): At 6-week, responsiveness (change in gait speed = 0.05 m/s) will be evaluated. Responders will continue with their assigned treatment and non-responders will be randomized to either continue assigned treatment or combined treatment for an additional 6 weeks.
  Interventions: Behavioral: Functional Power Training (FPT); Behavioral: Music-Based Digital Therapy (MBDT); Behavioral: FPT + MBDT

INTERVENTIONS:
Behavioral: Functional Power Training (FPT) — Participants will receive twice weekly FPT, a progressive functional-based exercises that target optimizing leg force production and leg velocity.
Behavioral: Music-Based Digital Therapy (MBDT) — Participants will receive twice weekly MBDT, a technology-driven gait training that is grounded in evidence-based rehabilitation treatment, rhythmic auditory stimulation.
Behavioral: FPT + MBDT — For non-responders who were randomized to augment treatment, they will receive combined FPT and MBDT treatment.
  Arms: Stage 2: Exercise Treatment

SUMMARY:
This study will begin to evaluate personalized preventative dementia treatments for Veterans at risk for developing dementia. The investigators will target Veterans with Motoric Cognitive Risk syndrome (MCR), which is characterized by slow gait speed and cognitive concerns (e.g., problems with memory or concentrations).

DETAILED DESCRIPTION:
This study will involve therapeutic exercise treatments for Veterans with pre-clinical dementia syndrome. Participants will either participate in functional power training, music-based walking training, or a combination of both. The study will use a sequential multiple assignment, randomized trial (SMART) design. Successful completion of this study will lay the foundation for subsequent research trials, contributing to valuable evidence for personalized rehabilitation medicine for older Veterans.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65
2. Receiving VA primary care
3. Community-dwelling
4. Motoric Cognitive Risky Syndrome i. Slow gait speed ii. Subjective cognitive concerns/complaints

Exclusion Criteria:

1. Non-English speaking
2. Presence of a terminal disease
3. Major medical problem
4. Myocardial infarction or major surgery in the previous 3 months
5. 3-point walking pattern
6. Dementia diagnostic
7. Mobility disability

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment/Baseline | Enrollment
  Enrollment will be defined as the number of participants who were recruited and consented to the study.
Retention | Baseline to end of 12-week treatment
  Retention will be defined as the number of participants who completed the 12-week exercise treatment.
Compliance | Baseline to end of 12-week treatment
  Compliance will be defined by the proportion of completed treatment sessions.
Acceptability | End of 12-week treatment
  Acceptability will be recorded by conducting interviews with participants who completed the 12-week exercise treatment.

SECONDARY OUTCOMES:
Gait Speed | Baseline to end of 12-week treatment
  Change in gait speed will be assessed after 12-week exercise treatment.

OTHER OUTCOMES:
Cognition - Executive Function | Baseline to end of 12-week treatment
  Change in executive function will be assessed after 12-week exercise treatment using Delis-Kaplan Executive Function System.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Ogawa, PhD MS BS, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No